CLINICAL TRIAL: NCT04687735
Title: Minimally Invasive Technique to Increase the Range of Motion of the Shoulder Joint in Frozen Shoulder: Single Arm Prospective Study
Brief Title: Frozen Shoulder Single Arm Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allevio Pain Management Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2357-3002-5
Record Dates: First submitted 2020-12-03; First posted 2020-12-29 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-01

CONDITIONS: Frozen Shoulder
Keywords: Brachial Plexus Block; Physical Therapy; Quality of Life
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: single-center, prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Patients with frozen shoulders at any stage
  Interventions: Other: Intervention after nerve block

INTERVENTIONS:
Other: Intervention after nerve block — Brachial plexus block + Physical therapy

SUMMARY:
The purpose of this study is to evaluate the effect of combination of brachial plexus block plus physical therapy on quality of life improvement in patients with frozen shoulder condition via standard questionnaires.

DETAILED DESCRIPTION:
STUDY OBJECTIVES The primary objective is to evaluate the effect of combination of regional anesthesia and physical therapy measured as an improvement in pain related disability scores of the impaired shoulder using the Shoulder Disability Questionnaire (SDQ), Shoulder Pain and Disability Index (SPADI), and improvement in pain score measured by Brief Pain Inventory (BPI).

The secondary objectives are to evaluate the effect of treatment on the following:

* Anxiety, measured by General Anxiety Disorder Questionnaire (GAD-7)
* Depression, measured by Beck's Depression Inventory (BDI)
* Satisfaction, measured by Global Improvement and Satisfaction Score (GISS) STUDY DESIGN This is as a single-center, prospective cohort study. The study does not imply any new intervention; all decisions regarding the treatment will be made at the sole discretion of the treating physician as part of clinical care. The study will be conducted over a period of 14 months, including approximately 1-2 months of enrolment, 4-6 weeks of treatment and follow-up at 3, 6, 12 months after the initiation of treatment for frozen shoulder. Treatment 1 can be scheduled along with baseline consult and screening (Day 0), three to five more treatment visits (Treatment 2 to Treatment 6) will be scheduled weekly (4-6 treatments in total), and follow up visits on 3, 6, and 12 months (with ±1week window). If patient has achieved any early full ROM, treatment will be stopped according to the physicians' decision. The study will be conducted at the Allevio Pain Clinic, Toronto, Canada. Research Ethics approvals will be sought.

STUDY POPULATION Patients with unilateral or bilateral frozen shoulder in any stage will be screened for study eligibility.

STUDY INTERVENTION

1st part of treatment: (by Anesthesiologist) Treatment will be provided to all eligible patients at baseline visit (Day 0). In the procedure room, after exposing the affected shoulder, the skin of the shoulder and neck on the affected area will be be prepared with the mixture of chlorhexidine and alcohol. The position of the patient will be decided based on the preference of the practitioner for performing brachial plexus block. Some of our practitioners prefer to perform the procedure on supine position and some prefer lateral position. Any difference in performing the brachial plexus block on supine or lateral position is not expected. Furthermore, using a familiar position for the anesthesiologist performing the brachial plexus block only adds to the safety of the intervention.

The anesthesiologist will use ultrasound and a sterile technique to perform two procedures:

* In the first step, with the guidance of ultrasound, brachial plexus block (inter scalene approach) will be provided. In total, 10 mL of a very dilute local anesthetic, marcaine 0.08 %, would be injected. The real-time guidance of ultrasound will be used to monitor the whole procedure. By using an ultrasound guidance, the practitioner wiill make sure that the local anesthetic has reached to all three nerve roots in inter scalene space.
* In the second step of the procedure, the patient will be asked to sit up. In this step, normal saline will be injected into the shoulder joint. The posterior approach will be used with the real-time guidance of ultrasound. Depending on the compliance of the shoulder joint, between 10-40 mL of normal saline will be injected. The target area for normal saline is between the shoulder capsule and the head of the humorous. The goal is to use the hydrostatic pressure to lift the capsule and separate the layers of adhesion from the cartilage of the head of humorous.

The patient will stay in the recovery area for 15 minutes after both interventions are performed. For the entire duration of both procedures, pulse rate, blood pressure, and oxygen saturation in the room air will continuously be monitored every 5 minutes. Then the patient will be moved to another area of the clinic to start physical therapy.

Physical therapy:

On the consult plus treatment day, assessment of the shoulder will begin in the seated position. The range of passive external rotation will be measured with the elbow held tight to the torso and bent at 90 degrees. Care will be taken to ensure that the patient does not rotate at the trunk during external rotation of the shoulder. Manual palpation of the coracoid process and deltoid insertion will be performed to check for pain and/or point sensitivity.

The patient then will be placed in the supine position to check passive flexion and abduction of the shoulder. Care will be taken to ensure the patient does not hike the shoulder towards the ear during the passive abduction or arch the back during passive flexion, thereby allowing evaluation solely of the rotator cuff. Due to the relatively small sample size and working within a very active clinic environment, a visual estimation of the passive ROM will be recorded in 20-degree increments.

After physical assessment and suitability confirmation, patients will be scheduled for 4-6 treatment appointments where they will undergo brachial plexus block and shoulder joint injection by the anesthesiologist before passive mobilization performed by the chiropractor. Each passive mobilization treatment will be generally 20 minutes in duration. Care will be directed solely at the affected shoulder, and no other passive modalities will be applied other than manual mobilization. The patient will be given three home based exercises to perform. These exercises are pendulums, passive external rotation against a door frame, and active wall walks within the patient's pain tolerance. The patient will be asked to perform 2 sets of exercises once a day, at 10 repetitions per set.

STUDY VISITS AND PROCEDURES Study visits and related procedures are displayed in Table 1. During the screening visit the study coordinator will obtain informed consent and perform eligibility check, (which has been explained in recruitment section). Additional visits may be required to address patient questions and to sign informed consent, collect demographics (age, gender, race), medical history, clinical data. Qualified participants will be scheduled for their combined appointment with anesthesiologist and chiropractor at the same time (Baseline visit), and thereafter every week for 4-6 weeks depend on ROM achievement.

On the baseline visit, after routine documentation of the blood pressure, heart rate and saturation of oxygen in room air and completion of baseline questionnaires, the patient would move to the procedure room to receive the intervention that is described above.

Questionnaires will also be collected at each follow-up visits. Furthermore, the investigator will perform the following procedures at all visits:

* perform clinical examination,
* report adverse events (AE) and/or serious adverse events (SAE), and
* complete relevant section of case report form (CRF)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of unilateral or bilateral frozen shoulder, defined as greater than 50% limitation of passive ROM relative to the non affected side in one or more of three movement directions (i.e., abduction in the frontal plane, forward flexion in the sagittal plane, or external rotation in 0° of abduction) with a hard end feel
* Symptoms of frozen shoulder that had lasted for at least 3 months.
* Willing and able to provide informed consent and perform home-based exercises as instructed.
* Willing and able to complete study questionnaires

Exclusion Criteria:

* Previous manipulation of the affected shoulder under anesthesia in the last year;
* Other rheumatic conditions involving the shoulder (e.g., rheumatoid arthritis, ankylosing Spondylitis,
* Fracture or dislocation of the affected shoulder;
* Previous shoulder surgery;
* Hill-Sachs lesion, severe osteoporosis, or malignancies in the shoulder region);
* Neurologic deficits affecting shoulder function;
* History of allergy to lidocaine;
* Corticosteroid injection in the affected shoulder during the receding 4 weeks.
* Non-English speakers;
* Active non- controlled mental disorders
* Multiple complete tear in ligaments of rotator cuff
* Any infection including COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
changes in disability score | 12 months
  measured by Shoulder Disability Questionnaire (descriptive format No= no disability, Yes= disable)
changes in disability score | 12 months
  measured by Shoulder Pain and Disability Index, min 0, max 10, 0 means no pain and disability and 10 means the worst pain and disability

SECONDARY OUTCOMES:
Changes in pain score (If there is any pain) | 12 months
  measured by short form of Brief Pain Inventory Questionnaire min 0, max 10, 0 means no pain and disability and 10 means the worst pain and disability
Changes in anxiety score | 12 months
  measured by General Anxiety Disorder Questionnaire min 0, max 21, 0 means no anxiety and 21 means the maximum anxiety
Changes in depression score | 12 months
  measured by Beck's Depression Inventory min 0, max 40, 0 means no depression and 40 means the sever depression
Changes in treatment satisfaction | 12 months
  using the Global Improvement and Satisfaction Score, between 1 to 5, 1 very dissatisfied, and 5 very satisfied
Frequency and duration of treatment related side | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Allevio Pain Management, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pal B, Anderson J, Dick WC, Griffiths ID. Limitation of joint mobility and shoulder capsulitis in insulin- and non-insulin-dependent diabetes mellitus. Br J Rheumatol. 1986 May;25(2):147-51. doi: 10.1093/rheumatology/25.2.147. PMID 3708230
- [Result] Uppal HS, Evans JP, Smith C. Frozen shoulder: A systematic review of therapeutic options. World J Orthop. 2015 Mar 18;6(2):263-8. doi: 10.5312/wjo.v6.i2.263. eCollection 2015 Mar 18. PMID 25793166
- [Result] Hand GC, Athanasou NA, Matthews T, Carr AJ. The pathology of frozen shoulder. J Bone Joint Surg Br. 2007 Jul;89(7):928-32. doi: 10.1302/0301-620X.89B7.19097. PMID 17673588
- [Result] Rodeo SA, Hannafin JA, Tom J, Warren RF, Wickiewicz TL. Immunolocalization of cytokines and their receptors in adhesive capsulitis of the shoulder. J Orthop Res. 1997 May;15(3):427-36. doi: 10.1002/jor.1100150316. PMID 9246090
- [Result] Tamai K, Akutsu M, Yano Y. Primary frozen shoulder: brief review of pathology and imaging abnormalities. J Orthop Sci. 2014 Jan;19(1):1-5. doi: 10.1007/s00776-013-0495-x. Epub 2013 Dec 4. PMID 24306579
- [Result] Riddle DL, Rothstein JM, Lamb RL. Goniometric reliability in a clinical setting. Shoulder measurements. Phys Ther. 1987 May;67(5):668-73. doi: 10.1093/ptj/67.5.668. PMID 3575423
- [Result] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Result] Homsi C, Bordalo-Rodrigues M, da Silva JJ, Stump XM. Ultrasound in adhesive capsulitis of the shoulder: is assessment of the coracohumeral ligament a valuable diagnostic tool? Skeletal Radiol. 2006 Sep;35(9):673-8. doi: 10.1007/s00256-006-0136-y. Epub 2006 May 25. PMID 16724200
- [Result] Ando A, Hamada J, Hagiwara Y, Sekiguchi T, Koide M, Itoi E. Short-term Clinical Results of Manipulation Under Ultrasound-Guided Brachial Plexus Block in Patients with Idiopathic Frozen Shoulder and Diabetic Secondary Frozen Shoulder. Open Orthop J. 2018 Mar 16;12:99-104. doi: 10.2174/1874325001812010099. eCollection 2018. PMID 29619123
- [Result] YAMSHON LJ. Frozen shoulder: methods for bringing about early mobilization. Calif Med. 1958 Nov;89(5):333-4. PMID 13585158
- [Result] Hsu WC, Wang TL, Lin YJ, Hsieh LF, Tsai CM, Huang KH. Addition of lidocaine injection immediately before physiotherapy for frozen shoulder: a randomized controlled trial. PLoS One. 2015 Feb 25;10(2):e0118217. doi: 10.1371/journal.pone.0118217. eCollection 2015. PMID 25714415
- [Result] Kanbe K. Clinical outcome of arthroscopic capsular release for frozen shoulder: essential technical points in 255 patients. J Orthop Surg Res. 2018 Mar 16;13(1):56. doi: 10.1186/s13018-018-0758-5. PMID 29548325
- [Result] Paul A, Rajkumar JS, Peter S, Lambert L. Effectiveness of sustained stretching of the inferior capsule in the management of a frozen shoulder. Clin Orthop Relat Res. 2014 Jul;472(7):2262-8. doi: 10.1007/s11999-014-3581-2. Epub 2014 Mar 25. PMID 24664198
- [Result] Rymaruk S, Peach C. Indications for hydrodilatation for frozen shoulder. EFORT Open Rev. 2017 Nov 22;2(11):462-468. doi: 10.1302/2058-5241.2.160061. eCollection 2017 Nov. PMID 29218231
- [Result] Maund E, Craig D, Suekarran S, Neilson A, Wright K, Brealey S, Dennis L, Goodchild L, Hanchard N, Rangan A, Richardson G, Robertson J, McDaid C. Management of frozen shoulder: a systematic review and cost-effectiveness analysis. Health Technol Assess. 2012;16(11):1-264. doi: 10.3310/hta16110. PMID 22405512
- [Result] Lewis J. Frozen shoulder contracture syndrome - Aetiology, diagnosis and management. Man Ther. 2015 Feb;20(1):2-9. doi: 10.1016/j.math.2014.07.006. Epub 2014 Jul 18. PMID 25107826
- [Result] Rookmoneea M, Dennis L, Brealey S, Rangan A, White B, McDaid C, Harden M. The effectiveness of interventions in the management of patients with primary frozen shoulder. J Bone Joint Surg Br. 2010 Sep;92(9):1267-72. doi: 10.1302/0301-620X.92B9.24282. PMID 20798446
- [Result] Vastamaki H, Varjonen L, Vastamaki M. Optimal time for manipulation of frozen shoulder may be between 6 and 9 months. Scand J Surg. 2015 Dec;104(4):260-6. doi: 10.1177/1457496914566637. Epub 2015 Jan 26. PMID 25623916
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171